CLINICAL TRIAL: NCT04128917
Title: A Randomized, Double-Blind, Active-controlled, Multicenter, Pilot Study to Investigate the Safety and Efficacy of a Triple Therapy With Tegoprazan, Amoxicillin and Clarithromycin in H. Pylori Positive Patients
Brief Title: Triple Therapy With Tegoprazan in H. Pylori Positive Patients_PILOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_E01
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50 mg (Experimental): Tegoprazan 50 mg Triple Therapy
  Interventions: Drug: Tegoprazan
- Tegoprazan 100 mg (Experimental): Tegoprazan 100 mg Triple Therapy
  Interventions: Drug: Tegoprazan
- RAPAE01 (Active Comparator): RAPAE01 Triple Therapy
  Interventions: Drug: RAPAE01

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg or 100 mg/Clarithromycin/Amoxicillin BID peroral
  Arms: Tegoprazan 100 mg; Tegoprazan 50 mg
Drug: RAPAE01 — RAPAE01/Clarithromycin/Amoxicillin BID peroral
  Arms: RAPAE01

SUMMARY:
This study aims to compare safety and efficacy in an exploratory manner between a Tegoprazan triple therapy and a RAPAE01 triple therapy in H. pylori positive patients.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Active-controlled, Multicenter, Pilot Study to Investigate the Safety and Efficacy of a Tegoprazan triple therapy and a RAPAE01 triple therapy in H. pylori positive patients.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori positive at screening
* Subjects who have upper gastrointestinal disease

Exclusion Criteria:

* Having received prior therapy for eradication of H. pylori
* Prior use of P-CAB, proton pump inhibitors (PPIs), H2 receptor blockers within 14 days
* Prior use of H. pylori eradication effective antibiotics, bismuth within 28 days

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | Day 49
  Assess H. pylori eradication rate by UBT

CONTACTS AND LOCATIONS:
Overall Officials: JAEGYU KIM, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JY, Choi IJ, Kim GH, Hong SJ, Shin SK, Jeon SW, Kim JG. Comparative Efficacy of Potassium-Competitive Acid Blocker-Based Triple Therapy with Tegoprazan versus Vonoprazan for Helicobacter pylori Eradication: A Randomized, Double-Blind, Active-Controlled Pilot Study. Gut Liver. 2025 Sep 15;19(5):696-705. doi: 10.5009/gnl250067. Epub 2025 Jun 4. PMID 40462641